CLINICAL TRIAL: NCT05387759
Title: A Randomized, Double-blind, Placebo- and Positive-controlled, Single-dose, 4-way Crossover Study to Evaluate the Effects of Aticaprant (JNJ-67953964) on Electrocardiogram Intervals in Healthy Adult Participants
Brief Title: A Thorough QT Study of Aticaprant (JNJ-67953964) in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CR109186; 2021-002618-15 (EudraCT Number); 67953964MDD1001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2022-05-20; First posted 2022-05-24 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Healthy
MeSH Terms: interventions — Aticaprant; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Treatment Sequence 1 (Experimental): Healthy participants will receive single oral dose of Aticaprant (Dose 1) (Treatment A) in Treatment Period 1, followed by Moxifloxacin (Dose 2) (Treatment D) in Treatment Period 2, followed by Aticaprant (Dose 3) (Treatment B) in Treatment Period 3 and then placebo (Treatment C) in Treatment Period 4, on Day 1 of each treatment period. There will be a wash-out period up to 7-15 days between each treatment period.
  Interventions: Drug: Aticaprant Supratherapeutic Dose; Drug: Aticaprant Therapeutic Dose; Drug: Placebo; Drug: Moxifloxacin
- Treatment Sequence 2 (Experimental): Healthy participants will receive single oral dose of Treatment B in Treatment Period 1, followed by Treatment A in Treatment Period 2, followed by Treatment C in Treatment Period 3 and then Treatment D in Treatment Period 4, on Day 1 of each treatment period. There will be a wash-out period up to 7-15 days between each treatment period.
  Interventions: Drug: Aticaprant Supratherapeutic Dose; Drug: Aticaprant Therapeutic Dose; Drug: Placebo; Drug: Moxifloxacin
- Treatment Sequence 3 (Experimental): Healthy participants will receive single oral dose of Treatment C in Treatment Period 1, followed by Treatment B in Treatment Period 2, followed by Treatment D in Treatment Period 3 and then Treatment A in Treatment Period 4, on Day 1 of each treatment period. There will be a wash-out period up to 7-15 days between each treatment period.
  Interventions: Drug: Aticaprant Supratherapeutic Dose; Drug: Aticaprant Therapeutic Dose; Drug: Placebo; Drug: Moxifloxacin
- Treatment Sequence 4 (Experimental): Healthy participants will receive single oral dose of Treatment D in Treatment Period 1, followed by Treatment C in Treatment Period 2, followed by Treatment A in Treatment Period 3 and then Treatment B in Treatment Period 4, on Day 1 of each treatment period. There will be a wash-out period up to 7 to 15 days between each treatment period.
  Interventions: Drug: Aticaprant Supratherapeutic Dose; Drug: Aticaprant Therapeutic Dose; Drug: Placebo; Drug: Moxifloxacin

INTERVENTIONS:
Drug: Aticaprant Supratherapeutic Dose — Aticaprant supratherapeutic dose capsule will be administered orally.
  Other Names: JNJ-67953964
Drug: Aticaprant Therapeutic Dose — Aticaprant therapeutic dose capsule will be administered orally.
  Other Names: JNJ-67953964
Drug: Placebo — Placebo will be administered orally.
Drug: Moxifloxacin — Moxifloxacin capsule will be administered orally.

SUMMARY:
The purpose of this study is to assess the effects of aticaprant on QT/ QT interval corrected for heart rate (HR) (QTc) intervals and electrocardiogram (ECG) morphology at therapeutic and supratherapeutic exposures in healthy adult participants.

ELIGIBILITY:
Inclusion Criteria:

* Healthy on the basis of physical examination, medical history, vital signs, and 12-lead electrocardiogram (ECG) performed at screening and admission to the study center on Day -1 of the first treatment period. Minor abnormalities in ECG, which are not considered to be of clinical significance by the investigator, are acceptable
* Body mass index (BMI; weight [kilograms {kg}/ height square [meter square {m^2}]) between 18 and 30.0 kg/m^2 (inclusive), and body weight not less than 50 kg at screening
* All female participants must have a negative serum pregnancy test (Beta-human chorionic gonadotropin [Beta-hCG]) at screening and a negative urine pregnancy test at admission to the study site on Day -1 of the first treatment period
* A woman must agree not to donate eggs (ova, oocytes) or freeze for future use for the purposes of assisted reproduction during the study and for a period of at least 90 days after receiving the last dose of study intervention
* Non-smoker (not smoked for 3 months prior to screening)

Exclusion Criteria:

* History of or current significant medical illness including (but not limited to) cardiac arrhythmias or other cardiac disease, hematologic disease, lipid abnormalities, bronchospastic respiratory disease, diabetes mellitus, hepatic or renal insufficiency, thyroid disease, Parkinson's disease, infection, or any other illness that the investigator considers should exclude the participant
* History of additional risk factors for Torsade de Pointes or the presence of a family history of short QT syndrome, long QT syndrome, sudden unexplained death at a young age (less than/equal to 40 years), drowning or sudden infant death syndrome in a first degree relative (that is, biological parent, sibling, or child)
* Any skin condition likely to interfere with electrocardiographic electrode placement or adhesion
* Breast implant or a history of thoracic surgery likely to cause abnormality of the electrical conduction through thoracic tissues
* History of malignancy within 5 years before screening (exceptions are squamous and basal cell carcinomas of the skin and carcinoma in situ of the cervix, or malignancy, which is considered cured with minimal risk of recurrence)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-05-30 (Actual); Primary Completion 2022-10-04 (Actual); Study Completion 2022-10-04 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in QTc at Each Time Point | Baseline up to Day 4
  Change from baseline in QTc at each time point will be reported.

SECONDARY OUTCOMES:
Maximum Observed Concentration (Cmax) of Aticaprant | Predose up to 72 hours postdose (up to Day 4)
  Cmax is defined as the maximum observed plasma concentration of aticaprant and it's metabolite.
Time To Reach The Maximum Observed Concentration of Aticaprant (Tmax) | Predose up to 72 hours postdose (up to Day 4)
  Tmax is the actual sampling time to reach the maximum observed plasma concentration of aticaprant.
Area Under the Plasma Concentration-Time Curve From Time Zero to last of Aticaprant (AUC [0-last]) | Predose up to 72 hours postdose (up to Day 4)
  AUC (0-last) is the area under the plasma concentration-time curve from time 0 to the time of the last measurable (non-below quantification limit) concentration of aticaprant.
Area Under the Plasma Concentration-Time Curve From Time Zero to Infinite Time of Aticaprant (AUC[0-infinity]) | Predose up to 72 hours postdose (up to Day 4)
  AUC (0-infinity) is the area under the plasma concentration-time curve from time zero to infinite time of aticaprant.
Number of Participants With Adverse Events (AEs) | Up to Day 4
  Number of participants with AEs will be reported. An AE is any untoward medical occurrence in a clinical study participant administered a pharmaceutical (investigational or non investigational) product.
Number of Participants with AEs of Special Interest (AESI) | Up to Day 4
  Number of participants with AESIs will be reported. Pruritus and severe diarrhea is considered to be an AESI.
Number of Participants With Change in Vital Signs | Up to Day 4
  Number of participants with change in vital signs will be reported. Body temperature, blood pressure, and pulse/heart rate (HR) measurements will be assessed.
Number of Participants With Change in Laboratory Values | Up to Day 4
  Number of participants with change in laboratory parameters will be reported. Hematology, serum chemistry, and routine urinalysis will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Clinical Pharmacology Unit, Merksem, Belgium

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency